CLINICAL TRIAL: NCT02212691
Title: Functional Neuroimaging of Pain in Sickle Cell Disease Patients
Brief Title: Functional Neuroimaging of Pain Using EEG and fMRI
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1211M24481; U01HL117664 (NIH)
Record Dates: First submitted 2014-08-01; First posted 2014-08-08 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Sickle cell disease: Patients diagnosed with sickle cell disease
- Healthy control: Healthy individuals recruited through fliers and have no history of cognitive disorders

SUMMARY:
The purpose of this research is to use non-invasive imaging technologies to study how the human brain processes pain. The investigators will use contact heat to induce pain and record data scalp EEG and functional magnetic resonance imaging (fMRI). What the investigators learn from this study will help us gain insights in pain management with broad socioeconomic impacts

DETAILED DESCRIPTION:
Functional imaging of brain networks associated with pain processing is of vital importance to aid developing new pain-relief therapy and to better understand the mechanisms of brain function. The pain response in the brain is a complex process, which involves multiple cortical brain regions, such as primary and secondary somatosensory cortices, anterior cingulate cortex, and insular cortex . Recent advancement in neuroimaging techniques suggests the possibility to map the brain structure and networks that involve pain processing. Electroencephalography (EEG) is a noninvasive monitoring technique, which is widely used to probe neurological disorders with high temporal resolution. Few attempts have been made to use EEG to map the active brain regions in pain patients. Functional MRI (fMRI) measures the hemodynamic brain response and could image the active brain regions with high spatial resolution. Studies have shown that fMRI is a useful tool to delineate the brain regions associated with pain processing. Recent studies from simultaneous EEG and fMRI recording have suggested that the EEG response to the pain may be correlated with the fMRI response, and both EEG and fMRI could be used to image the brain pain processing regions, such as the primary somatosensory cortex and anterior cingulate cortex.

The aim of this research is to develop and evaluate a functional neuroimaging approach using EEG, fMRI and EEG-fMRI, in pain study. EEG, fMRI, or simultaneous EEG-fMRI will be collected in healthy subjects who receive external thermal stimulation inducing pain. The painful stimuli will be delivered at different intensity levels and the subject pain rating will be collected. The imaging technique combines the EEG signal with high temporal resolution and the fMRI signal with high spatial resolution to obtain a spatiotemporal imaging of the brain electrophysiological and hemodynamic activity in response to different levels of pain. Cross validation between this method and subject pain score will be used to quantitatively and qualitatively evaluate the technique. The successful completion of the current protocol will help establish an important imaging technology accessing pain level in an objective way.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects with no known neurological disorders
* Sickle cell patients with no metal implants

Exclusion Criteria:

* Age over 65 in either group

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy subjects Sickle cell patients
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2012-01; Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Changes in EEG power | up to four years
  The goal is to find biomarkers using EEG/fMRI to noninvasively quantify pain. The investigators will measure the differences in EEG power in patients with sickle cell disease comparing to healthy controls.
Changes in fMRI activity level | up to four years
  The goal is to find biomarkers using EEG/fMRI to noninvasively quantify pain. The investigators will measure the differences in fMRI BOLD activation in patients with sickle cell disease comparing to healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Bin He, PhD, Principal Investigator — University of Minnesota
Locations (1):
- Biomedical Engineering Department, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Case M, Shirinpour S, Zhang H, Datta YH, Nelson SC, Sadak KT, Gupta K, He B. Increased theta band EEG power in sickle cell disease patients. J Pain Res. 2017 Dec 27;11:67-76. doi: 10.2147/JPR.S145581. eCollection 2018. PMID 29343982
- [Result] Case M, Shirinpour S, Vijayakumar V, Zhang H, Datta Y, Nelson S, Pergami P, Darbari DS, Gupta K, He B. Graph theory analysis reveals how sickle cell disease impacts neural networks of patients with more severe disease. Neuroimage Clin. 2019;21:101599. doi: 10.1016/j.nicl.2018.11.009. Epub 2018 Nov 14. PMID 30477765

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-28): https://cdn.clinicaltrials.gov/large-docs/91/NCT02212691/Prot_SAP_000.pdf